CLINICAL TRIAL: NCT04316260
Title: Development and Testing of a Smoking Cessation E-Visit for Implementation in Primary Care
Brief Title: Smoking Cessation E-Visit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jennifer Dahne, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00078077
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking cessation electronic visit (e-visit) (Experimental): This group will be sent 1) an invitation to complete an electronic visit (e-visit) focused on cigarette smoking and 2) an invitation to complete a follow-up e-visit one-month after the initial e-visit.
  Interventions: Behavioral: Smoking cessation e-visit
- Treatment As Usual (Active Comparator): This group will be provided information about the state quitline and about the importance of quitting smoking and it will be recommended that they contact their PCP to schedule a medical visit to discuss quitting smoking.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Smoking cessation e-visit — electronic visits (e-visits) for smoking cessation
  Arms: Smoking cessation electronic visit (e-visit)
Behavioral: Treatment As Usual — Information about the state quitline and about the importance of quitting smoking and a recommendation to contact one's PCP to schedule a medical visit to discuss quitting smoking
  Arms: Treatment As Usual

SUMMARY:
The goal of this study is to develop, refine, and complete preliminary feasibility testing of a smoking cessation electronic visit (e-visit) for implementation in primary care/family medicine. The investigators will conduct a feasibility RCT (N=51) of the smoking cessation e-visit as compared to treatment as usual (TAU), delivered via primary care, with primary objective to provide effect size estimates for a larger RCT. Primary outcomes cluster around: 1) treatment feasibility, 2) treatment acceptability, 3) treatment satisfaction, 4) evidence-based cessation treatment utilization, and 5) cessation-related outcomes (quit attempt incidence, abstinence). It is hypothesized that participants randomized to the e-visit condition as compared to those randomized to the TAU condition will have higher rates of cessation treatment utilization (medications, counseling) and superior cessation-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. current smoking, defined as smoking 5+ cigarettes/day, for 20+ days out of the last 30, for the last 6+ months
2. age 18+
3. enrolled in Epic's MyChart program or willing to sign up for MyChart
4. possess a valid e-mail address that is checked daily to access follow-up assessments and MyChart messages
5. English fluency

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dahne J, Player M, Carpenter MJ, Ford DW, Diaz VA. Evaluation of a Proactive Smoking Cessation Electronic Visit to Extend the Reach of Evidence-Based Cessation Treatment via Primary Care. Telemed J E Health. 2021 Mar;27(3):347-354. doi: 10.1089/tmj.2020.0167. Epub 2020 Oct 20. PMID 33085578

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Started | 34 | 17
Completed | 34 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual | Total
Number analyzed (Participants) | 34 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.21 (13.42) | 42.76 (11.22) | 46.39 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 12 | 35
  Male | 11 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 33 | 17 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 6 | 17
  White | 22 | 8 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 34 | 17 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Utilized Smoking Cessation Treatment
Description: Number of participants who utilized smoking cessation treatment since last assessment.
Time Frame: Month 1
Population: The number of participants analyzed differs from the total participants in each group because not everyone completed the questionnaire that assessed this information.
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Number analyzed (Participants) | 28 | 17
Participants | 15 | 3

2. Primary Outcome: Number of Participants Who Utilized Smoking Cessation Treatment
Description: Number of participants who utilized smoking cessation treatment since last assessment.
Time Frame: Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Number analyzed (Participants) | 23 | 16
Participants | 14 | 4

3. Secondary Outcome: E-visit Completion
Description: Number of participants that completed the e-visit
Time Frame: Month 1
Measure: Count of Participants; unit: Participants
Groups:
- Smoking Cessation E-visit (Electronic Visit) Group: This group will be sent 1) an invitation to complete an electronic visit (e-visit) focused on cigarette smoking and 2) an invitation to complete a follow-up e-visit one-month after the initial e-visit.
  Smoking cessation e-visit: electronic visits (e-visits) for smoking cessation
Arm/Group | Smoking Cessation E-visit (Electronic Visit) Group
Number analyzed (Participants) | 34
Participants | 19

4. Primary Outcome: Cigarettes Smoking
Description: Cigarettes per day reduction greater than 50%
Time Frame: Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Number analyzed (Participants) | 28 | 17
Participants | 9 | 3

5. Primary Outcome: Cigarettes Smoking
Description: Cigarettes per day reduction greater than 50%
Time Frame: Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Number analyzed (Participants) | 23 | 16
Participants | 15 | 5

6. Primary Outcome: Quit Attempts
Description: Quit attempts since last contact
Time Frame: Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Number analyzed (Participants) | 28 | 17
Participants | 16 | 5

7. Primary Outcome: Quit Attempts
Description: Quit attempts since last contact
Time Frame: Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Number analyzed (Participants) | 23 | 16
Participants | 14 | 12

8. Primary Outcome: 24-hour Quit Attempt
Description: Quit attempt lasting 24 hours since last contact
Time Frame: Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Number analyzed (Participants) | 28 | 17
Participants | 11 | 4

9. Primary Outcome: 24-hour Quit Attempt
Description: Quit attempt lasting 24 hours since last contact
Time Frame: Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Number analyzed (Participants) | 23 | 16
Participants | 11 | 11

10. Primary Outcome: Seven-day Point Prevalence Abstinence
Description: Participant has not had a cigarette in the past 7 days
Time Frame: Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Number analyzed (Participants) | 28 | 17
Participants | 3 | 0

11. Primary Outcome: Seven-day Point Prevalence Abstinence
Description: Participant has not had a cigarette in the past 7 days
Time Frame: Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Number analyzed (Participants) | 23 | 16
Participants | 5 | 1

12. Primary Outcome: Floating Abstinence
Description: Participant has gone 7+ days without a cigarette since last contact.
Time Frame: Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Number analyzed (Participants) | 28 | 17
Participants | 4 | 1

13. Primary Outcome: Floating Abstinence
Description: Participant has gone 7+ days without a cigarette since last contact.
Time Frame: Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
Number analyzed (Participants) | 23 | 16
Participants | 7 | 4

14. Secondary Outcome: Provider Fidelity
Description: Reviewing within Epic whether the provider administered treatment consistent with e-visit recommendations
Time Frame: Month 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation E-visit (Electronic Visit) Group
Number analyzed (Participants) | 34
Participants | 27

15. Secondary Outcome: E-visit Ease of Use
Description: Participants reported Agree or Strongly Agree to finding the e-visit easy to use question
Time Frame: Month 1
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation E-visit (Electronic Visit) Group
Number analyzed (Participants) | 34
Participants | 25

16. Secondary Outcome: Time to Complete the E-visit
Description: Time (days) to complete the e-visit among participants that completed the e-visit.
Time Frame: Month 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Smoking Cessation E-visit (Electronic Visit) Group
Number analyzed (Participants) | 19
days | 1.42 (2.27)

ADVERSE EVENTS:
Time Frame: 1 month and 3 month assessments (3 total months)
Arm/Group | Smoking Cessation Electronic Visit (E-visit) | Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/17
Other Adverse Events (participants affected / at risk) | 4/34 | 3/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smoking Cessation Electronic Visit (E-visit) (N=34) | Treatment As Usual (N=17)
Headaches (Nervous system disorders) | 2 (3) | 2 (3)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Insomnia/trouble sleeping (Psychiatric disorders) | 2 (3) | 2 (4)
Nausea (Nervous system disorders) | 1 (1) | 1 (1)
Sleep problems (Psychiatric disorders) | 2 (2) | 3 (4)
Depressed mood (Psychiatric disorders) | 2 (3) | 1 (2)
Appetite change (Gastrointestinal disorders) | 1 (1) | 1 (1)
Weight loss/gain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Agitation/hostility (Social circumstances) | 2 (2) | 2 (2)
Heartburn (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ringing in the ears (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT04316260/Prot_SAP_000.pdf